CLINICAL TRIAL: NCT01718626
Title: Study Comparing Sequential Therapy of S1+Docetaxel Followed by S1 to Concomitant S1+Docetaxel for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hebei Tumor Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBTH101
Record Dates: First submitted 2012-10-25; First posted 2012-10-31 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

ARMS (2):
- S1+Docetaxel (Active Comparator)
  Interventions: Drug: S1+Docetaxel
- S1+Docetaxel followed by S1 (Experimental)
  Interventions: Drug: S1+Docetaxel followed by S1

INTERVENTIONS:
Drug: S1+Docetaxel — Drug: S1 40-60mg, bid, days1-14, every 3 weeks Docetaxel 50mg/m2, day1, every 3 weeks, Patients will receive S1+Docetaxel until progression
  Arms: S1+Docetaxel
Drug: S1+Docetaxel followed by S1 — Drug: S1 40-60mg, bid, days1-14, every 3 weeks Docetaxel 50mg/m2, day1, every 3 weeks,for 4 cycles; S1 40-60mg, bid, days1-14, every 3 weeks Patients will receive S1+Docetaxel followed by S1 until progression
  Arms: S1+Docetaxel followed by S1

SUMMARY:
Stage 1:First line therapy Sequential therapy of S1+Docetaxel followed by S1 is superior to concomitant S1+Docetaxel in the safety and clinical efficiency.

Stage 2:Second line therapy To explore the feasibility of single drug(S1) maintenance treatment for advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Performance Status-Eastern Cooperative Oncology Group (ECOG) 0-1
* Histologically or cytologically confirmed gastric cancer
* Advanced or recurrent, metastatic disease
* At least have one measurable disease(according to RECIST, Response Evaluation Criteria in Solid Tumors )
* Life expectancy of at least 3 months
* Target target lesion has not received radiotherapy or non target lesion radiation at least 4 weeks
* Haematopoietic and Hepatic status:

Absolute neutrophil count >1.5x109/L,Platelet count > 100 x 109/L,Hemoglobin at least 9 g/dl,Bilirubin ≤ 1.5 x upper limit of normal (ULN),AST and ALT ≤ 2.5 times ULN(no liver metastasis), ≤5 times ULN(with liver metastasis)

* Cardiovascular: Baseline LVEF 50% measured by echocardiography

Exclusion Criteria:

* Symptomatic brain metastasis
* Active or uncontrolled infection
* Unresolved or unstable, serious toxicity from prior cancer treatment (any toxicities greater than grade 2; peripheral neuropathy of grade 2 or greater Symptomatic brain metastasis
* Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, uncontrolled hypertension (≥ 180/110), unstable diabetes mellitus, dyspnea at rest, or chronic therapy with oxygen
* History of other malignancy
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 1 years

SECONDARY OUTCOMES:
Objective response rate(ORR) | 1 year
Disease control rate(DCR) | 1 year
Overall survival(OS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Wei Liu, Principal Investigator — Hebei Tumor Hospital
Locations (1):
- Department of Medical Oncology, Shijiazhuang, Hebei, China